CLINICAL TRIAL: NCT00891267
Title: Effect of Olmesartan Medoxomil on Vascular Markers in Hypertensive Patients With Metabolic Syndrome
Brief Title: Effect of Two Doses of Olmesartan Medoxomil and Amlodipine on Vascular Markers in Hypertensive Patients With Metabolic Syndrome
Acronym: VAMOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo Europe, GmbH, a Daiichi Sankyo Company (Industry)
Responsible Party: Senior Manager Clinical Development, Daiichi Sankyo Europe
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: DSE-866/46; 2007-003130-41 EudraCT number
Record Dates: First submitted 2009-04-29; First posted 2009-05-01 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2011-05

CONDITIONS: Metabolic Syndrome; Hypertension
Keywords: Inflammatory markers; Vascular protection; OM Effect; Metabolic syndrome; Hypertension
MeSH Terms: conditions — Metabolic Syndrome; Hypertension | interventions — Olmesartan Medoxomil; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Olmesartan medoxomil low dose (Experimental): Olmesartan medoxomil tablets low dose, taken once daily for 6 weeks
  Interventions: Drug: Olmesartan medoxomil tablets low dose
- Olmesartan medoxomil tablets high dose (Experimental): Olmesartan medoxomil tablets high dose, taken once daily for 6 weeks
  Interventions: Drug: Olmesartan medoxomil tablets high dose
- Amlodipine (Active Comparator): Amlodipine taken once daily for 6 weeks
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Olmesartan medoxomil tablets low dose — Olmesartan medoxomil tablets low dose, taken once daily for 6 weeks
  Arms: Olmesartan medoxomil low dose
Drug: Olmesartan medoxomil tablets high dose — Olmesartan medoxomil tablets high dose, taken once daily for 6 weeks
  Arms: Olmesartan medoxomil tablets high dose
Drug: Amlodipine — Amlodipine tablets taken once daily for 6 weeks
  Arms: Amlodipine

SUMMARY:
The purpose of this study is to study the effect of two doses of olmesartan medoxomil and amlodipine on vascular markers in hypertensive patients with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Male and female Europeans at the age of 18 years or above with hypertension, metabolic syndrome, and modest inflammation
* Blood pressure greater than or equal to 130/85 mmHg AND
* hs-CRP greater than or equal to 1.0 and less than 10.0 mg/dL AND at least two (2) of the following traits of the metabolic syndrome (ATP III criteria):
* abdominal obesity: waist circumference greater than 102 cm for men and 88 cm for women;
* triglyceride level greater than or equal to 150 mg/dL; HDL less than 40 mg/dL for men and less than 50 mg/dL for women
* fasting blood glucose greater than or equal to 110mg/dL

Exclusion Criteria:

* Insulin depended diabetes or type-1 diabetes
* Severe or resistant hypertension
* Patients with secondary hypertension of any aetiology, such as renal disease, pheochromocytoma, or Cushing's syndrome
* Any acute or chronic inflammatory disease
* Constant use of lipid-lowering agents (eg statins, fibrates) for less than 3 months before study start
* Pregnant or lactating female patients of childbearing potential (prerequisite: adequate contraception);
* Patients with serious disorders which may limit the ability to evaluate the efficacy or safety of the trial drug(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-10; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To investigate the anti-inflammatory effect of Olmesartan (OM) higher dose compared to Olmesartan (OM) lower dose and amlodipine (AML) on the change in levels of the inflammatory marker hs-CRP | 6 weeks for each treatment

SECONDARY OUTCOMES:
To evaluate the additional antihypertensive efficacy in blood pressure (BP) lowering, assessed by conventional BP measurement and 24-h ambulatory BP measurement (24-h ABPM) | 6 weeks for each treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Erlangen, Germany

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/